CLINICAL TRIAL: NCT01454323
Title: Phase II Clinical Trial on the Effect of Intracoronary Infusion of Bone Marrow Mononuclear Cells on Functional Recovery in Patients With Myocardial Chronic Back and Severely Depressed Left Ventricular Function.
Brief Title: Intracoronary Infusion of Bone Marrow Mononuclear Cells in Patients With Previous Myocardial Infarction.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMMo/CIC/2009; 2009-016599-66 (EudraCT Number)
Record Dates: First submitted 2011-10-12; First posted 2011-10-19 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Myocardial Ischemia
Keywords: Chronic Myocardial Ischemia; Cell therapy; Bone marrow mononuclear cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Dose of bone marrow mononuclear cells: 5-7 x 108 total cells
  Interventions: Other: Bone marrow mononuclear cells

INTERVENTIONS:
Other: Bone marrow mononuclear cells — Intracoronary infusion of autologous bone marrow-derived mononuclear cells

SUMMARY:
Phase II clinical trial which will include all patients diagnosed with chronic anterior myocardial infarction (more than 6 months from the acute phase and the complete revascularization in which it is assessed the evolution of left ventricular function in patients to the monitoring against their own basal condition.

Included patients will be studied in the following conditions:

* Basal condition: defined as the immediately preceding to the administration of cell therapy treatment.
* Monitoring Condition 1: three months after drug administration of cell therapy. Includes non-invasive methods of exploration of ventricular function.
* Monitoring Condition 2: six months after administration of treatment. Includes the same methods of exploration of ventricular function practised in the basal condition, including cardiac catheterism as well as non invasive methods.
* Monitoring Condition 3: twelve months after administration of the cell therapy drug. Includes non-invasive methods of exploration of ventricular function.

The trial hypothesis we propose consists of mononuclear cells of bone marrow providing progenitor cells with regenerative capacity and also secreting several angiogenic factors, and their implantation into ischemic tissues should contribute with both elements to the angiogenesis and tissue regeneration with myocardial functional recovery

DETAILED DESCRIPTION:
This is an uncontrolled study in which the efficacy of the cell therapy drug is measured by comparing the variables of ventricular function after treatment to the basal condition prior to its application

The total number of patients to be studied 20. The study population will correspond to male and female patients with chronic anterior myocardial infarction (more than 6 months after the acute episode) and ventricular dysfunction. It is expected 36 months of inclusion and one year follow up

Patients will receive in a concomitant way the drug treatment established by the good practice, so it would certainly be possible that some improvement occurs due to drug treatment.

It will be studied the patient population of both genders aged between 18 and 80 years diagnosed with Chronic anterior myocardial infarction (more than 6 months after the acute phase and the complete revascularization).

Objectives of the study:

* Main objective: To determine the efficacy of intracoronary injection of adult stem cells from autologous bone marrow in patients with chronic anterior myocardial infarction in terms of improvement of ventricular function, determined by hemodynamic, echocardiographic and New York Heart Association (NYHA) functional class criteria, resulting in an improvement of heart failure symptoms and quality of life's patient.
* Secondary objectives:

  1. To investigate the basic cellular mechanisms underlying the myocardial regeneration process through correlation between hemodynamic criteria for the ventricular function improvement and the biologicals corresponding to the composition and the functionality of the infused cells.
  2. To analyze clinical, hemodynamic and biologicals factors able to influence favorably to a greater degree of functional recovery after regenerative treatment in chronic myocardial infarction.
  3. To design, in view of the results obtained, suitable protocol for the application of cell therapy to treat patients with old anterior infarction, both in terms of the ideal characteristics of medullary graft as in terms of those patients more likely to be beneficiaries of it, in order to establish a definitive strategy of including cell therapy in the standard treatment of this disease in the near future provided that the results indicate it so.

The primary variable is the improvement in ventricular function monitoring under angiographic and echocardiographic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years.
2. Patients diagnosed with Chronic anterior myocardial infarction (more than 6 months from the acute episode) with symptoms and / or signs of heart failure.
3. Left ventricular ejection fraction (LVEF)<45% and distensibility changes.
4. Complete revascularization performed at least 6 months before infusion cells.

Exclusion Criteria:

1. Patients in active waiting list for heart transplantation..
2. Treatable patients with resynchronization.
3. Patients over 80 years
4. Coexistence of other serious systemic diseases.
5. Active infection, HIV, Hepatitis B or Hepatitis C.
6. Patients with malignant or pre-malignant tumours.
7. Coexistence of any haematological disease.
8. Pregnant women, in breastfeeding period, or in childbearing potential age who are not using effective contraception.
9. Patients who are currently participating or have completed their participation in a clinical trial in a period of less than three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in left ventricular ejection fraction (LVEF) | 3, 6 and 12 months after intervention

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 12 months
Functional grade of the New York Heart Association (NYHA) | 3,6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Suarez de lezo, MD, PhD, Study Chair — University Hospital Reina Sofía, Córdoba.; Inmaculada Herrera, MD, PhD, Study Chair — University Hospital Reina Sofía, Córdoba.; Miguel Ángel Romero, MD, Principal Investigator — University Hospital Reina Sofía, Córdoba.
Locations (1):
- University Hospital Reina Sofía, Córdoba, Spain, Spain

REFERENCES:
- See also: Andalusian Molecular Biology and Regenerative Medicine Centre — http://www.cabimer.es